CLINICAL TRIAL: NCT01702090
Title: Early Access to TMC114 in Combination With Low-dose Ritonavir (TMC114/r) and Other Antiretrovirals (ARVs) for Treatment-naive or TMC114-naive, Early Treatment Experienced in HIV-1 Infected Patients
Brief Title: Early Access to Low-dose Ritonavir (TMC114/r) and Other Antiretrovirals (ARVs) for Treatment-naive or Early Treatment Experienced in HIV-1 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100712; TMC114HIV4073 (Other: Janssen-Cilag Ltd.); DRV-C-10-TW01-001 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2012-02-13; First posted 2012-10-05 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: HIV-1
Keywords: HIV-1; TMC114; Darunavir; PREZISTA; Ritonavir; Antiretrovirals; Early access; Early treatment; Treatment naive
MeSH Terms: interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMC114/ritonavir (Experimental)
  Interventions: Drug: TMC114/ritonavir

INTERVENTIONS:
Drug: TMC114/ritonavir — TMC114 800 mg (two tablets) once daily coadministered with ritonavir 100 mg (one capsule) once daily within 30 minutes after completion of a meal, and in combination with other ARVs.
  Other Names: PI

SUMMARY:
The purpose of this study is to provide early access to TMC114 administered with low-dose ritonavir (TMC114/r) and other antiretrovirals (ARVs) for HIV-1-infected patients who have not received previous HIV treatment or have received early treatment without TMC114 regimens.

DETAILED DESCRIPTION:
This is a single-treatment-group, open-label (patients and study personnel will know the identity of the treatments given), single-center study. The primary goal of this study is to provide early access to TMC114 administered with low-dose ritonavir (TMC114/r) and other antiretrovirals (ARVs, agents that are used to treat viral infections). This study is intended for HIV-1-infected patients who have not received previous HIV treatment (treatment-naive patients) or have received early treatment without TMC114 regimens and who are ineligible to participate in any other sponsored HIV-1 study. This study will monitor and evaluate the safety and efficacy of TMC114/r in combination with ARVs during the course of the study. Treatment with TMC114/r will be continued until virologic failure (the inability to achieve or maintain suppression of viral replication), treatment-limiting toxicity, loss to follow-up, study withdrawal, pregnancy, until discontinuation of TMC114 development or when TMC114 becomes reimbursable for treatment-naive patients or when TMC114 becomes commercially available for treatment-experienced patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HIV-1 infection who are ineligible for participation in any other Sponsor's HIV-1 trial
* Patients have never been treated with antiretroviral (ARV) medications or have prior early treatment-experienced without TMC114 regimens, including they have limited or no treatment options due to virological failure or intolerance to regimens
* Patient's general medical condition, in the investigator's opinion evaluating the patient is eligible for TMC114 containing regimen, does not interfere with the assessments and the completion of the trial

Exclusion Criteria:

* Any active clinically significant disease or findings during screening of medical history or physical examination that is not either resolved or stabilized for at least 30 days before the screening phase of the trial
* Evidence of active liver disease, acute viral hepatitis, liver impairment/dysfunction or cirrhosis irrespective of liver enzyme levels; however, patients coinfected with hepatitis B or C will be included if their condition is judged to be clinically stable
* Grade 3 or 4 laboratory abnormalities as defined by Division of AIDS (DAIDS).
* Calculated creatinine clearance (CrCl) less than 50 ml/min
* Female patients that are pregnant or breast-feeding, or of childbearing potential without using effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last 30 days after the end of the treatment period
* Any condition (including but not limited to alcohol and/or drug abuse), which in the opinion of the investigator, could compromise the patient's safety or compliance to the study protocol procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma HIV-1 RNA level | Day 1 (Baseline) up to end-of-study visit, an expected average of approximately 3 months
  End-of-study visit is defined as the time TMC114 becomes commercially available or reimbursed for treatment-naïve patients.
Change in plasma CD4 cell count | Day 1 (Baseline) up to end-of-study visit, an expected average of approximately 3 months
  End-of-study visit is defined as the time TMC114 becomes commercially available or reimbursed for treatment-naïve patients.

SECONDARY OUTCOMES:
Number of participants affected by an adverse event | Up to end-of-study visit, an expected average of approximately 3 months
  End-of-study visit is defined as the time TMC114 becomes commercially available or reimbursed for treatment-naïve patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, MD and PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Taipei, Taiwan

REFERENCES:
- See also: Early access to TMC114 in combination with low-dose ritonavir (tmc114/r) and other Antiretrovirals (AVRs) for treatment-naïve or TMC114-naïve, early treatment-experienced in HIV-1 infected patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3374&filename=CR100712_CSR.pdf